CLINICAL TRIAL: NCT06088524
Title: Determining the Effects of Mental Fatigue Created by Social Media on Upper Extremity Performance
Brief Title: The Effects of Mental Fatigue Created by Social Media on Upper Extremity Performance
Status: Completed | Type: Observational
Sponsor: Bandırma Onyedi Eylül University (Other)
Collaborators: Burçin Akçay (Unknown); Arzu Genç (Unknown); Canan Demir (Unknown)
Responsible Party: Principal Investigator, Ozan Bahadır Turkmen, PhD Candidate, Bandırma Onyedi Eylül University
Other Study IDs: 2022-187
Record Dates: First submitted 2023-09-12; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Mental Fatigue; Upper Extremity Performance; Social Media
MeSH Terms: conditions — Mental Fatigue

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Social Media Fatigue — Mental Fatigue creation protocol: It has been reported that at least 30 minutes of social media use causes mental fatigue and impairs lower extremity and decision-making performance (Fortes et al., 2021). For mental fatigue with social media, participants will be created with 45 minutes of continuous use of social media (instagram, facebook, twitter, youtube) on smartphones by concentrating with headphones.

SUMMARY:
There are a limited number of studies in the literature, and it is stated that mental fatigue caused by social media use causes a decrease in upper-extremity movement speed and a decrease in lower-extremity endurance performance. Therefore, this study aims to determine the effects of social media-induced mental fatigue on upper extremity performance.

DETAILED DESCRIPTION:
Mental fatigue is a psychobiological condition that requires prolonged cognitive activity and is characterized by subjective feelings of "tiredness" and "lack of energy." It reduces sport-related decision-making, technical skills, motor control and endurance performances. This has led to a condition known as social media fatigue among many users, where they feel exhausted from repeated exposure to an enormous amount of information from brands. Social media fatigue is "the tendency of social media users to withdraw from social media when they are overwhelmed by too many social media sites, too many friends and followers, and too much time spent online to maintain these connections".Researchers have drawn attention to the negative effects of internet-induced fatigue, which is increasing daily, and emphasized that excessive internet use can lead to physical and psychological problems. Although there are a limited number of studies in the literature, there is a limited number of studies investigating the effects of mental fatigue caused by social media use on upper extremity performance.Therefore, this study aims to determine the effects of mental fatigue caused by social media on upper extremity performance.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Being sedentary
* To be between the ages of 18-30

Exclusion Criteria:

* Any mental or sensory problems in the last six months
* Acute infection or chronic disease of neurological, psychiatric, orthopedic, cardiological, rheumatological, etc. origin
* Having had any upper extremity injury and/or operation (trauma, surgery, fracture, etc.) in the last six months
* Regular medication use

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: It will be conducted on Bandırma Onyedi Eylül University Faculty of Health Sciences students.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
1-Isometric Elbow Flexion Strength | Baseline
  The participant will sit in a chair with upper arms at their sides, elbow bent 90 degrees, and forearm supinated. A velcro strap attached to a digital dynamometer fixed to a portable wooden platform placed under the chair will be secured tightly around the participant's wrist, proximal to the distal wrist crease. The tester will check the strap's tension to ensure no slack. When instructed, the participant will endeavor to move their hand as forcefully as possible towards the shoulder for 2-3 seconds. Any compensatory movement in trunk extension or lateral flexion outside the tested arm will be observed.
1-Isometric Elbow Flexion Strength | 1 week later
  The participant will sit in a chair with upper arms at their sides, elbow bent 90 degrees, and forearm supinated. A velcro strap attached to a digital dynamometer fixed to a portable wooden platform placed under the chair will be secured tightly around the participant's wrist, proximal to the distal wrist crease. The tester will check the strap's tension to ensure no slack. When instructed, the participant will endeavor to move their hand as forcefully as possible towards the shoulder for 2-3 seconds. Any compensatory movement in trunk extension or lateral flexion outside the tested arm will be observed.
2-Hand grip strength | Baseline
  Hand grip strength will be assessed using a Jamar hand dynamometer (Lafayette Instrument Company, USA). The participant will sit holding the dynamometer with the upper arm at the side, elbow bent 90 degrees, and forearm centered between pronation and supination. When instructed, the participant will squeeze the dynamometer as forcefully as possible for 2-3 seconds while the tester verbally encourages.
2-Hand grip strength | 1 week later
  Hand grip strength will be assessed using a Jamar hand dynamometer (Lafayette Instrument Company, USA). The participant will sit holding the dynamometer with the upper arm at the side, elbow bent 90 degrees, and forearm centered between pronation and supination. When instructed, the participant will squeeze the dynamometer as forcefully as possible for 2-3 seconds while the tester verbally encourages.
3- Upper extremity reaction test | Baseline
  It is planned to use the BlazePod sensor, validated for the upper extremity reaction time test (de-Oliveira et al. 2021).
3- Upper extremity reaction test | 1 week later
  It is planned to use the BlazePod sensor, validated for the upper extremity reaction time test (de-Oliveira et al. 2021).
4-Finger reaction test | Baseline
  The participant will be asked to place the dominant hand's index finger on the left button of a computer mouse and press the left button as soon as the green lights up on the traffic light shape on the screen. The time between the light stimulus and the participant's reaction will be recorded in milliseconds.
4-Finger reaction test | 1 week later
  The participant will be asked to place the dominant hand's index finger on the left button of a computer mouse and press the left button as soon as the green lights up on the traffic light shape on the screen. The time between the light stimulus and the participant's reaction will be recorded in milliseconds.
5-Hand performance test | Baseline
  The nine-hole peg test will be used. The 9-hole peg test (9-DPT) is a validated method widely used in research and clinical settings as a measure of finger dexterity (Y. A. Smith, Hong, & Presson, 2000).
5-Hand performance test | 1 week later
  The nine-hole peg test will be used. The 9-hole peg test (9-DPT) is a validated method widely used in research and clinical settings as a measure of finger dexterity (Y. A. Smith, Hong, & Presson, 2000).
6-Mental stopwatch | Baseline
  The Nine Hole Peg Test (9-DPT) was used to assess the temporal correspondence between actual and imagined movement. The 9-DPT will be administered according to standard protocols. The participant performed the test according to the standard 9-DPT protocol, during which the stopwatch will be started, and the time from the beginning to the end of the test will be recorded. In the imagined 9-DPT, a mental stopwatch will be used, and the same test will be performed with the individual visualizing the same activity while sitting with his/her eyes closed (Allali, 2012).
6-Mental stopwatch | 1 week later
  The Nine Hole Peg Test (9-DPT) was used to assess the temporal correspondence between actual and imagined movement. The 9-DPT will be administered according to standard protocols. The participant performed the test according to the standard 9-DPT protocol, during which the stopwatch will be started, and the time from the beginning to the end of the test will be recorded. In the imagined 9-DPT, a mental stopwatch will be used, and the same test will be performed with the individual visualizing the same activity while sitting with his/her eyes closed (Allali, 2012).
7-Evaluation of position sense | Baseline
  In the study, a Baseline® digital goniometer with a sensitivity of 1° will be used to assess the glenohumeral joint position sense. The tested person will be asked to perform shoulder flexion at 55°, 90° and 125° and to lift the arm from the position adjacent to the body to the angles mentioned (Balke et al., 2011).
7-Evaluation of position sense | 1 week later
  In the study, a Baseline® digital goniometer with a sensitivity of 1° will be used to assess the glenohumeral joint position sense. The tested person will be asked to perform shoulder flexion at 55°, 90° and 125° and to lift the arm from the position adjacent to the body to the angles mentioned (Balke et al., 2011).
8-Upper extremity endurance test: | Baseline
  After weighing the body weight, the weight in the hand will be calculated as 2% of the body weight and rounded to the nearest 0.5 kg if it is fractional. The participant will hang from the bed with his/her arm out. He/she should then take the weight in his/her hand and lift it with the "thumb pointing upwards" and the arm at 90° to the horizontal. A metronome set to 60 Hz will then be used to standardize the test, whereby participants will be instructed to raise their arm on the first beat, hold it at 90 abductions for the next beat and then lower it to the starting position on the third beat. The test will be terminated by fulfilling any of the following termination criteria (Moore, Uhl, & Kibler, 2013).
8-Upper extremity endurance test: | 1 week later
  After weighing the body weight, the weight in the hand will be calculated as 2% of the body weight and rounded to the nearest 0.5 kg if it is fractional. The participant will hang from the bed with his/her arm out. He/she should then take the weight in his/her hand and lift it with the "thumb pointing upwards" and the arm at 90° to the horizontal. A metronome set to 60 Hz will then be used to standardize the test, whereby participants will be instructed to raise their arm on the first beat, hold it at 90 abductions for the next beat and then lower it to the starting position on the third beat. The test will be terminated by fulfilling any of the following termination criteria (Moore, Uhl, & Kibler, 2013).

CONTACTS AND LOCATIONS:
Locations (1):
- Bandirma Onyedi Eylul University, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No